CLINICAL TRIAL: NCT03029000
Title: A Single-Arm Study of the Effect of a 5-day Regimen of Tbo-Filgrastim 10 mcg/kg of Body Weight Administered Subcutaneously on Peripheral Stem Cell Mobilization in Healthy Donors
Brief Title: Study of the Effect of a 5-Day Regimen of Study Drug on Peripheral Stem Cell Mobilization in Healthy Participants
Acronym: GRANIX
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to low enrollment
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV44688-ONC-30054
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tbo-filgrastim (GRANIX) (Experimental): Participants will receive tbo-filgrastim 10 mcg/kg of body weight, subcutaneously on the morning of Days 1 to 5.
  The actual dose of tbo-filgrastim administered to each, individual participant will be calculated at baseline according to his or her body weight and that specific dose (10 mcg/kg of body weight) for each, individual participant will remain the same for all consecutive daily doses.
  If the collection goal will not meet after the first apheresis on Day 5, tbo-filgrastim 10 mcg/kg of body weight will be administered subcutaneously for up to 3 additional days (Days 6 to 8) followed by daily apheresis to reach the cumulative collection goal.
  Interventions: Drug: Tbo-filgrastim

INTERVENTIONS:
Drug: Tbo-filgrastim — solution for subcutaneous injection
  Other Names: XM02

SUMMARY:
A multi-center, open-label, single-arm clinical study to assess effects of a 5-day regimen of 10 micrograms per kilogram (mcg/kg) of tbo-filgrastim administered subcutaneously daily on the mobilization of cluster of differentiation 34+ (CD34+) cells in at least 60 healthy male and female participants. The pharmacokinetics, pharmacodynamics, safety, tolerability, and immunogenicity of tbo-filgrastim will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained from the participant
* The participant has a body weight of at least 50 kilograms (kg)
* The participant has a body mass index (BMI) of more than 18.5 and less than 35.0 kilograms per square meter (kg/m^2)
* The participant is in good health as determined by medical and psychiatric history, physical examination, electrocardiogram (ECG) recordings, serum chemistry, hematology, coagulation, urinalysis, and serology
* Women may be included only if they have a negative beta human chorionic gonadotropin (beta-hCG) test at baseline, are sterile (defined as documented hysterectomy, bilateral oophorectomy or bilateral salpingectomy, or congenitally sterile), or postmenopausal (defined as no menses for 12 months without alternative medical cause and increased follicle stimulating hormone [FSH] of above 35 units per liter [U/L] in women not using hormonal contraception or hormonal replacement therapy). Women of childbearing potential whose male partners are potentially fertile (that is, no vasectomy) must use highly effective birth control methods for the duration of the study and for 30 days after the last tbo-filgrastim administration
* The participant has a negative alcohol urine test and a negative urine drug screen
* The participant must be willing and able to comply with study restrictions
* The participant is human leukocyte antigen (HLA) -matched or haploidentical-related to the recipient

Exclusion Criteria:

* The participant currently has or had a history of any clinically relevant gastrointestinal, hematologic, respiratory, psychiatric, renal, hepatic, cardiac, metabolic (such as, fructose intolerance), neurological, or any other disease or condition which may influence the physiological metabolic turnover (such as, severe endocrine diseases, febrile condition, severe infections), which may interfere with the study objectives, or which could expose the participant to undue risk through the participation in the clinical study
* The participant has had: (1) a trauma or surgery in the past 2 months; (2) a clinically relevant illness within 4 weeks before the first dose of tbo-filgrastim; (3) any acute illness within 1 week before the first dose of tbo-filgrastim; or (4) symptoms of any clinically relevant or acute illness at baseline
* The participant has existence or recent history of persistent pulmonary infiltrates, recent pneumonia, recent bronchitis, recurrent lung infections, or history or evidence of any lung disease including asthma, or current symptoms of upper respiratory tract infection. In the case of pneumonia, participant may be screened 12 weeks after cessation of antibiotic treatment
* The participant has findings of splenomegaly on sonography at screening, defined by length of spleen more than 12.3 centimeters (cm) and clinical judgment
* The participant has a history of malignancy, including hematologic malignancy, except for appropriately treated non-melanoma skin carcinoma in the last 5 years
* The participant has a clinically significant deviation from normal in ECG recordings or physical examination findings, as determined by the investigator
* The participant is pregnant or lactating, or was pregnant in the previous 6 months, or intends to get pregnant during the study or within 30 days after the last dose of study drug
* The participant has habitually consumed, within the last 2 years, more than 21 units of alcohol per week, or has a history or evidence of alcohol, narcotic, or any other substance abuse as defined by the Diagnostic and Statistical Manual of Mental Disorder, Fifth Edition (DSM-V, American Psychiatric Association 2013). Note: A unit of alcohol is equal to 1 ounce (29.6 milliliters [mL]) of hard liquor, 5 ounces (148 mL) of wine, or 8 ounces (236.8 mL) of beer
* The participant has taken any of the following investigational medicinal products (IMPs), medicinal products, or substances:

  1. Any IMP within 30 days or 5 half-lives (whichever is longer) before the first dose of tbo-filgrastim, or in the case of a new chemical entity, 3 months or 5 half-lives (whichever is longer) before the first dose of tbo-filgrastim
  2. Known history of treatment with blood-cell colony-stimulating factors
  3. Current or recent (within 4 weeks) treatment with lithium
* The participant has donated plasma within 7 days before screening or has donated blood within 56 days before screening
* The participant has a documented or self-reported history of tuberculosis or recent travel to countries of endemic disease (last 8 weeks)
* The participant has 1 or more clinical laboratory test value(s) outside the range specified below, or any other clinically significant laboratory abnormality as determined by the investigator or medical monitor:

  1. Hemoglobin less than or equal to (<=) 12.5 grams per deciliter (g/dL) (women) and hemoglobin <=13.5 g/dL (men)
  2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values of greater than (>) 3 * the upper limit of the normal range (ULN)
  3. Total bilirubin of >2 * ULN
  4. Findings of cholestasis (eg, abnormal values of alkaline phosphatase)
* The participant has a positive test result for human immunodeficiency virus (HIV), hepatitis B surface antigen, antibodies to hepatitis C virus, immunoglobulin M (IgM) antibodies to cytomegalovirus, human T-lymphotropic virus, West Nile virus, malaria, or syphilis
* The participant has a documented or self-reported history of tuberculosis or recent travel to countries of endemic disease (last 8 weeks)
* The participant has, after resting for 5 minutes, increased blood pressure (BP) (defined as systolic BP in seated position of more than 145 millimeters of mercury [mm Hg] or diastolic BP in seated position of more than 95 mm Hg), or low BP (defined as systolic BP in seated position of less than 90 mm Hg or diastolic BP in seated position of less than 45 mm Hg) (Only 2 rechecks of the participant's BP are permitted for eligibility purposes)
* The participant has, after resting for 5 minutes, a pulse in seated position of less than 45 or more than 90 beats per minute (Only 2 rechecks of the participant's pulse are permitted for eligibility purposes)
* The participant is unwilling to refrain from vigorous exercise (eg, strenuous or unaccustomed weight lifting, running, bicycling) from 72 hours before Day 1 until Day 15
* The participant is unlikely to comply with the study protocol or is unsuitable for any other reasons, as judged by the investigator
* The participant has a history of autoimmune disease, including rheumatic diseases and thyroid disorders
* The participant has a history of deep vein thrombosis or pulmonary embolism
* The participant has thrombocytopenia defined as platelet count <150 * 109 cells per liter (cells/L) at screening or at baseline
* The participant has a history of bleeding problems (eg, hemophilia, thrombocytopenia, idiopathic thrombocytopenic purpura, clotting factor deficiencies or disorders)
* The participant has positive hemoglobin-solubility test
* The participant has a history of iritis or episcleritis
* The participant has a history of significant hypersensitivity, intolerance, or allergy to tbo-filgrastim or any other E. coli derived product or excipient, or other medicinal product, food, or substance, unless approved by the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (9):
- United States (9):
  - Teva Investigational Site 14029, Duarte, California
  - Teva Investigational Site 14025, La Jolla, California
  - Teva Investigational Site 14023, Beech Grove, Indiana
  - Teva Investigational Site 14026, Detroit, Michigan
  - Teva Investigational Site 14027, Chapel Hill, North Carolina
  - Teva Investigational Site 14030, Cincinnati, Ohio
  - Teva Investigational Site 14033, Greenville, South Carolina
  - Teva Investigational Site 14035, Memphis, Tennessee
  - Teva Investigational Site 14024, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 6 participants were screened for this study, of which 5 participants were considered a screen failure mainly due to inclusion criteria not met or exclusion criteria met. Only one participant was enrolled and treated in this study.
Groups:
- Tbo-Filgrastim (GRANIX): Participant received tbo-filgrastim 10 micrograms per kilogram (mcg/kg) of body weight, administered subcutaneously on the morning of Days 1 to 5.
Period: Overall Study
Arm/Group | Tbo-Filgrastim (GRANIX)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled donor participants, regardless of whether or not a participant was administered tbo-filgrastim.
Groups:
- Tbo-Filgrastim (GRANIX): Participant received tbo-filgrastim 10 mcg/kg of body weight, administered subcutaneously on the morning of Days 1 to 5.
Arm/Group | Tbo-Filgrastim (GRANIX)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 2*10^6 Cluster of Differentiation 34+ (CD34+) Cells Per Kilogram (Cells/kg) of Recipient Body Weight Collected in the First Apheresis on Day 5
Description: The measurement of CD34+ cells in the apheresis product was performed by the local laboratory according to institutional guidelines.
Time Frame: Day 5
Population: Participants who received 5-day regimen of tbo-filgrastim 10 mcg/kg of body weight; and for whom, Day 5 apheresis was performed as planned and a quantifiable count of CD34+ cells in blood collected in Day 5 apheresis was measured.
Measure: Number; unit: percentage of participants
Arm/Group | Tbo-Filgrastim (GRANIX)
Number analyzed (Participants) | 1
percentage of participants | 100

2. Secondary Outcome: Percentage of Participants With at Least 2*10^6 CD34+ Cells/kg of Donor Baseline Body Weight Collected After the First Apheresis on Day 5
Description: as for outcome 1
Time Frame: Day 5
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Tbo-Filgrastim (GRANIX)
Number analyzed (Participants) | 1
percentage of participants | 100

3. Secondary Outcome: Percentage of Participants With at Least 5*10^6 CD34+ Cells/kg of Recipient Body Weight Collected After the First Apheresis on Day 5
Description: as for outcome 1
Time Frame: Day 5
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Tbo-Filgrastim (GRANIX)
Number analyzed (Participants) | 1
percentage of participants | 100

4. Secondary Outcome: Number of Aphereses Necessary to Collect at Least 5*10^6 CD34+ Cells/kg of Recipient Body Weight
Description: as for outcome 1
Time Frame: Days 5 to 8
Population: as for outcome 1
Measure: Number; unit: aphereses
Arm/Group | Tbo-Filgrastim (GRANIX)
Number analyzed (Participants) | 1
aphereses | 1

5. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs presented here included both SAEs and non-serious AEs.
Time Frame: From first administration of study drug (Day 1) up to early termination/end of study (up to approximately 3 months)
Population: Safety analysis set included all participants who received at least 1 dose of tbo-filgrastim.
Measure: Number; unit: percentage of particicpants
Arm/Group | Tbo-Filgrastim (GRANIX)
Number analyzed (Participants) | 1
percentage of particicpants | 100

6. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA)
Description: Blood samples (5 milliliters [mL]) for analysis of ADA were obtained for all participants at timepoints described.
Time Frame: Baseline (Day -3) up to early termination/end of study (up to approximately 3 months)
Population: Safety analysis set included all participants who received at least 1 dose of tbo-filgrastim.
Measure: Number; unit: percentage of participants
Arm/Group | Tbo-Filgrastim (GRANIX)
Number analyzed (Participants) | 1
percentage of participants | 0

7. Secondary Outcome: Maximum Observed Serum Recombinant Methionyl Human Granulocyte Colony-Stimulating Factor (r-metHuG-CSF) Concentration (Cmax)
Description: Blood samples were drawn for all participants for the determination of serum r-metHuG-CSF concentrations on Day 4. Pharmacokinetic (PK) parameter was calculated from concentration-time data using non compartmental methods, when possible.
Time Frame: Day 4 (8 hours post-dose)
Population: PK analysis set included all participants who received at least 1 dose of tbo-filgrastim and had at least 1 calculated PK parameter for tbo-filgrastim.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Tbo-Filgrastim (GRANIX)
Number analyzed (Participants) | 1
picograms per milliliter (pg/mL) | 19912.8

8. Secondary Outcome: Maximum Observed Peripheral CD34+ Cell Count (CD34+Cmax)
Description: Serial blood samples for the determination of CD34+ cell count were drawn.
Time Frame: Between Day 1 (pre-dose) and before the first apheresis on Day 5
Population: Pharmacodynamic (PD) analysis set included all participants who received at least 1 dose of tbo-filgrastim and had at least 1 calculated PD parameter.
Measure: Number; unit: cells per microliter (cells/mcL)
Arm/Group | Tbo-Filgrastim (GRANIX)
Number analyzed (Participants) | 1
cells per microliter (cells/mcL) | 144

ADVERSE EVENTS:
Time Frame: From first administration of study drug (Day 1) up to early termination/end of study (up to approximately 3 months)
Description: Safety analysis set included all participants who received at least 1 dose of tbo-filgrastim.
Arm/Group | Tbo-Filgrastim (GRANIX)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tbo-Filgrastim (GRANIX) (N=1)
Pain (General disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to operational feasibility. The decision to terminate the study was not related to any new or emerging safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT03029000/Prot_SAP_000.pdf